CLINICAL TRIAL: NCT04138693
Title: A Randomized, Placebo-controlled, Double-blind Study to Evaluate the Effect of G-PUR® on Enteral Lead Isotope 204Pb-absorption
Brief Title: G-PUR® for Reduced Lead Bioavailability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glock Health, Science and Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G-Lead_01
Record Dates: First submitted 2019-10-16; First posted 2019-10-24 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Lead Exposure
Keywords: Blood/Urine/Hair lead; Lead uptake & Lead bioavailability

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: 2 x 2.0 g G-PUR® oral suspension (Experimental)
  Interventions: Device: G-PUR® 2x 2.0 g oral suspension
- Cohort 2: 1 x 2.0 g G-PUR® oral suspension (Experimental)
  Interventions: Device: G-PUR® 1x 2.0 g oral suspension
- Cohort 3: Placebo oral suspension (Placebo Comparator)
  Interventions: Device: Placebo oral suspension

INTERVENTIONS:
Device: G-PUR® 2x 2.0 g oral suspension — Cohort 1: 2 g G-PUR® powder mixed with 100 ml water in an opaque drinking bottle will be orally administered before and immediately after 204Pb intake
  Arms: Cohort 1: 2 x 2.0 g G-PUR® oral suspension
Device: G-PUR® 1x 2.0 g oral suspension — Cohort 2: 2 g G-PUR® powder mixed with 100 ml water in an opaque drinking bottle will be orally administered before 204Pb intake and 100 ml water (placebo) in an opaque drinking bottle immediately after 204Pb intake
  Arms: Cohort 2: 1 x 2.0 g G-PUR® oral suspension
Device: Placebo oral suspension — Cohort 3: 100 ml of water in an opaque drinking bottle will be orally administered immediately before and after 204Pb intake
  Arms: Cohort 3: Placebo oral suspension

SUMMARY:
This is a prospective, randomized, placebo-controlled, double blind, parallel-arm study in a two-staged approach that will assess the effect of two different doses of G-PUR® on enteral lead absorption in healthy adults using a stable lead isotopic tracer (204Pb).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects
2. Age 18-45 years
3. BMI 19-27 for males and BMI 17-25 for female
4. Blood lead (PbB) concentration < 40 μg/l
5. Serum ferritin concentration within the sex-specific normal range, i.e. ≥ 15 - 150 ng/ml for women and 30 - 400 ng/ml for men
6. Presence of scalp hair with a minimum length of 5 mm and willingness to remove 5 single hairs with hair roots at end of study visit
7. Subject is in good clinical and mental health as established by medical history and physical examination
8. Stable eating habits, within one month before the start of the study
9. Subject agrees to be compliant for study related diet schedule
10. Women of childbearing potential agree to use adequate birth control methods during the study (for all females, negative pregnancy test at screening and at Visit 3 before dosing of IMD is required. Females of childbearing potential must use adequate contraception during the entire study period. Acceptable methods of contraception include: oral contraceptives, intrauterine device, female or male condoms with spermicide, diaphragm with spermicide, contraceptive medication patch, contraceptive medication implant, contraceptive medication injection, abstinence, or surgical sterilization more than 3 months before randomization.
11. Written informed consent

Exclusion Criteria:

1. Pregnancy and breastfeeding
2. Lack of willingness or capacity to co-operate appropriately
3. Regular use of medications or iron supplements in the previous 2 months except intake of contraceptives
4. Planning to shave head during study
5. History of malignancies within the past two years or on current anticancer treatment
6. History of gastrointestinal pathology such as gastritis, gastric ulcers, irritable bowel disease, inflammatory bowel disease, chronic constipation
7. History of diarrhoea within the past 14 days of screening
8. History of gastrointestinal surgery with exception of appendectomy
9. History of chronic autoimmune disease requiring treatment within the past two months of screening
10. Known diabetes mellitus I or II or Hba1c >6.5%
11. Known symptomatic food allergies
12. Any clinically relevant laboratory abnormalities in screening test
13. Alcohol, cigarette or drug abuse
14. Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
15. Presence of any condition that impacts compliance with the study procedures
16. Use of any regular medication (prescription or over the counter) for prevention or treatment of any medical condition
17. Use of any investigational or non-registered product (drug or device) within 30 days preceding the first study product administration, or planned use during the study period
18. Employee at the study site, spouse/partner or relative of any study staff (e.g. investigator, sub-investigators, or study nurse) or relationship to the sponsor
19. IMD should not be applied to patients that suffer from aluminium and/or silicon hypersensitivity or in case of renal failure that requires dialysis.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
204PbB Cmax normalized for total PbB | 216 hours
  Cmax of 204PbB normalized for total natural PbB levels after intake of 204Pb-enriched water

SECONDARY OUTCOMES:
Incidence of (S)ADE | 216 hours
  Incidence of (serious) adverse device effects
Plasma PK parameters - AUC0-t of 204PbB | 216 hours
  The observed area under the blood concentration versus time curve between time 0 and the time point of the last quantifiable concentration, calculated using the trapezoidal rule method
Plasma PK parameters - tmax of 204PbB | 216 hours
  Time to reach the peak concentration: The sampling time at which Cmax was observed
204Pb concentrations in 24-hour urine | 24 hours
  Measurement of 204Pb isotope tracer concentrations in 24-hour urine after intake of 204Pb enriched water
204Pb in single hairs | 9 days
  Lead isotope tracer (204Pb) distribution and ratio in single hairs

CONTACTS AND LOCATIONS:
Overall Officials: Christa Firbas, Dr., Principal Investigator — Medical University Vienna, Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Samekova K, Firbas C, Irrgeher J, Opper C, Prohaska T, Retzmann A, Tschegg C, Meisslitzer C, Tchaikovsky A, Gouya G, Freissmuth M, Wolzt M. Concomitant oral intake of purified clinoptilolite tuff (G-PUR) reduces enteral lead uptake in healthy humans. Sci Rep. 2021 Jul 20;11(1):14796. doi: 10.1038/s41598-021-94245-x. PMID 34285282